CLINICAL TRIAL: NCT02378415
Title: Subanesthetic IV Bolus Ketamine in the Treatment of Acute Depression
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Discrepancies in medication orders
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2011.0063
Record Dates: First submitted 2012-08-15; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Acute Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline Infusion (Placebo Comparator): A single IV bolus dose of normal saline solution.
  Interventions: Drug: Placebo
- Subanesthetic IV Bolus Ketamine (Experimental): a single sub-anesthetic rapid IV bolus dose of ketamine administered to acutely depressed patients with or without suicidality
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — IV Bolus dose of ketamine dosed at 0.2mg/kg infused over 1-2 minutes.
  Other Names: Ketalor.
  Arms: Subanesthetic IV Bolus Ketamine
Drug: Placebo — Normal Saline Infusion
  Arms: Normal Saline Infusion

SUMMARY:
The objective of this double-blinded placebo-controlled pilot study is to determine whether a single sub-anesthetic rapid IV bolus dose of ketamine administered to acutely depressed patients with or without suicidality has a significant rapid antidepressant effect in the acutely depressed population. The study will pursue as a primary outcome measure whether a significant reduction in depressive symptoms, as assessed by the BSS and BHS, occurs shortly after administration of ketamine at 40, 80, 120, and 240 minutes. A secondary outcome measure will be assessed to determine whether this single infusion of ketamine has a sustained reduction in depressive symptoms within 2-weeks post-infusion with a reduction in BDI score. Suicidal ideation will also be assessed for determination of any reduction and sustained reduction post infusion by assessment of the Beck Suicidal Ideation Scale (BSS), Beck Hopelessness Scale (BHS) and Beck Depression Inventory (BDI) at similar intervals.

DETAILED DESCRIPTION:
A determination for hospital admittance by a consulting psychiatrist will be made prior to study participation. Only those persons being admitted to the psychiatric ward will be eligible to enroll in this study. After consenting to participate in the trial and meeting inclusion criteria for this study (to include a baseline BDI, BSS, and BHS), voluntarily presenting acutely depressed patients, with or without suicidal ideation, will be randomized into two groups and administered standard of care treatment with intravenous ketamine (0.2mg/kg over 1-2 minutes) or standard of care treatment with intravenous normal saline (equal volume to ketamine dose). All prepared study solutions will be mixed and administered by ED staff and/or nursing staff as per the existing NMCSD ED protocols. All subjects will be blinded to the treatment given, either an IV bolus dose of ketamine at 0.2-mg/kg over 1-2 minutes or a placebo solution composed of an equal IV bolus dose (by overall volume) of 0.9 normal saline solution will be administered. Thereafter, all patients will be evaluated clinically with a BSS, BHS, and BDI at 40, 80, 120, and 240 minutes. All study participants will be monitored medically in the ED for at least the full 240-minute protocol and once declared medically clear, in accordance with standard of care practices by the ED providers, will be transferred to the inpatient psychiatric ward for further monitoring for at least 24-hours prior to discharge from the hospital. All enrolled patients will be administered another BSS, BHS, and BDI prior to discharge from the hospital. The length of hospital stay will also be recorded for further analysis, but will not be considered a secondary outcome measure for this study. Psychiatric determination for discharge from the hospital will be based on clinical assessment, presentation history, and hospital course and is not considered an outcome measure for this study. All patients included in this study will be re-assessed within 2 weeks with another BSS, BHS, and BDI for determination of sustainability of effects. Appropriate follow-up care with a psychiatrist will be afforded to all study participants after discharge from the hospital. Additionally, should any severe adverse side effects develop; the treatment administered to enrolled patients may be un-blinded by a third-party shift medical monitor (i.e. the Charge Nurse) on request from the emergency room provider. Additionally, given the potential psychotropic effects of ketamine and to assure that patients are sufficiently monitored and appropriately medically cleared, all participants in the study will be required to remain under clinical observation in the emergency room prior to transfer to the psychiatric ward for, at least, the full 4-hour treatment cycle or longer as clinically indicated. All participants in this study will only be allowed to enroll in this study and undergo this protocol's treatment once.

ELIGIBILITY:
Inclusion Criteria:

1. BSS greater than 4
2. BHS greater than 8
3. BDI greater than 19
4. Ability to give informed consent.
5. Active Duty military status.
6. Verified negative qualitative pregnancy test.
7. All participants must be accepted for psychiatric admission to the hospital PRIOR to consideration for enrollment in this study.

Exclusion Criteria:

1. Psychosis or Bipolar Disorder.
2. Pregnancy
3. Involuntary Status on presentation to the ED.
4. UDS positive for illicit drugs of abuse.
5. Blood Alcohol level greater than zero.
6. Previous enrollees in this treatment protocol will be excluded from repeat participation.
7. Any patient brought for command directed psychiatric evaluation.
8. Specific contraindications to the use of ketamine are as follows and under such circumstances or conditions, personnel with the following should be excluded from participation in this study:

   1. Patients with elevated intracranial pressure, uncontrolled hypertension, coronary artery disease, aneurysms, thyrotoxicosis, CHF, a recent history of head or eye injury, or angina.
   2. All personnel in whom a significant elevation of blood pressure would constitute a serious hazard to their overall health and well-being.
   3. Patients currently utilizing the following medications: conivaptan, Disatinib, peginterferon alfa-2b, quazepam, tocilizumab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Suicidality | Baseline
  Beck Suicidal Ideation Scale (BSS)

SECONDARY OUTCOMES:
Depression | Baseline, 40-minutes, 80-minutes, 120-minutes, 240-minutes, exit at discharge, and at follow-up within 2-weeks
  Beck Depression Index (BDI)
Hopelessness | Baseline, 40-minutes, 80-minutes, 120-minutes, 240-minutes, exit at discharge, and at follow-up within 2-weeks
  Beck Hopelessness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Lovern, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States